CLINICAL TRIAL: NCT06498778
Title: Prediction of Etiology and Prognosis Based on Hematoma Location of Spontaneous Intracerebral Hemorrhage
Brief Title: Etiology and Prognosis of sICH Based on Hemorrhage Location
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Guangming Lu, Director of the Medical Imaging Center of the Jinling Hospital, Jinling Hospital, China
Other Study IDs: 2022DZGZR-074
Record Dates: First submitted 2024-06-29; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Spontaneous Intracerebral Hemorrhage
Keywords: Normative analysis; Lesion-symptom mapping; Radiomics; Etiological classification; Machine learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- good outcome: Modified Rankin Scale (mRS) scores were determined based on clinical examinations or telephone follow-ups at twelve months post sICH event. Consistent with prior literature, we defined good outcome as "mRS = 0-2".
- poor outcome: Modified Rankin Scale (mRS) scores were determined based on clinical examinations or telephone follow-ups at twelve months post sICH event. Consistent with prior literature, we defined poor outcome as "mRS = 3-6".

SUMMARY:
The investigators retrospectively collected participants with spontaneous cerebral hemorrhage(sICH) from January 2015 to December 2019 for training and internal validation. Clinical and imaging data were collected. Modified Rankin Scale (mRS) scores were determined good outcome as "mRS = 0-2", poor outcome as "mRS = 3-6". The location features of sICH were extracted by symptom mapping. Noncontrast computed tomography images of patients and hematoma masks were registered with standard human brain templates to identify specific affected brain regions. Then a probability map of hemorrhage for different causes and prognosis is generated. PyRadiomics was used to extract the radiomic features, integrate radiomic and clinical features into multiple logistic regression models, and develop and validate optimal etiological and prognostic models. Further tests were performed in an independent cohort. The area under the working characteristic curve (AUC), sensibility, specificity were used to evaluate the reliability of the model.

ELIGIBILITY:
Inclusion Criteria:

* The confirmation of intracranial hemorrhage was achieved through NCCT.

Exclusion Criteria:

* They presented with secondary hemorrhage resulting from head trauma, hemorrhagic transformation of ischemic infarction, brain tumors, or exhibited abnormalities in blood coagulation, liver, kidney function, or were subject to drug-induced cerebral hemorrhage
* Only postoperative CT images were available
* Lost follow-up records
* CT image artifacts

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This retrospective study encompassed the collection of sICH patients. The confirmation of intracranial hemorrhage was achieved through NCCT.
Sampling Method: Probability Sample
Enrollment: 698 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) scores | follow-ups at twelve months post sICH event
  Good outcome as "mRS = 0-2", poor outcome as "mRS = 3-6"

CONTACTS AND LOCATIONS:
Overall Officials: Guangming Lu, Study Director — Deparetment of Radiology, Jinling Hospital
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Greenberg SM, Ziai WC, Cordonnier C, Dowlatshahi D, Francis B, Goldstein JN, Hemphill JC 3rd, Johnson R, Keigher KM, Mack WJ, Mocco J, Newton EJ, Ruff IM, Sansing LH, Schulman S, Selim MH, Sheth KN, Sprigg N, Sunnerhagen KS; American Heart Association/American Stroke Association. 2022 Guideline for the Management of Patients With Spontaneous Intracerebral Hemorrhage: A Guideline From the American Heart Association/American Stroke Association. Stroke. 2022 Jul;53(7):e282-e361. doi: 10.1161/STR.0000000000000407. Epub 2022 May 17. No abstract available. PMID 35579034
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Liu X, Zhang Q, Li J, Xu Q, Zhuo Z, Li J, Zhou X, Lu M, Zhou Q, Pan H, Wu N, Zhou Q, Shi F, Lu G, Liu Y, Zhang Z. Coordinatized lesion location analysis empowering ROI-based radiomics diagnosis on brain gliomas. Eur Radiol. 2023 Dec;33(12):8776-8787. doi: 10.1007/s00330-023-09871-y. Epub 2023 Jun 29. PMID 37382614
- [Background] Ding L, Liu H, Jing J, Jiang Y, Meng X, Chen Y, Zhao X, Niu H, Liu T, Wang Y, Li Z. Lesion Network Mapping for Neurological Deficit in Acute Ischemic Stroke. Ann Neurol. 2023 Sep;94(3):572-584. doi: 10.1002/ana.26721. Epub 2023 Jun 27. PMID 37314250
- [Background] Boe NJ, Hald SM, Jensen MM, Kristensen LMB, Bojsen JA, Elhakim MT, Clausen A, Moller S, Hallas J, Garcia Rodriguez LA, Selim M, Goldstein LB, Al-Shahi Salman R, Gaist D. Major Cardiovascular Events After Spontaneous Intracerebral Hemorrhage by Hematoma Location. JAMA Netw Open. 2023 Apr 3;6(4):e235882. doi: 10.1001/jamanetworkopen.2023.5882. PMID 37017964